CLINICAL TRIAL: NCT05338502
Title: An Open-Label, 3-Period, Fixed Sequence Study to Evaluate the Effect of an H2 Antagonist and a Proton Pump Inhibitor on the Single Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects
Brief Title: Study of H2 Antagonist and a Proton Pump Inhibitor of Selpercatinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17574; J2G-OX-JZJL (Other: Eli Lilly and Company); LOXO-RET-19075 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-04-19; First posted 2022-04-21 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib; Ranitidine; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 160 milligram (mg) Selpercatinib (Experimental): Participants received a single oral dose of 160 mg Selpercatinib (Study Day 1).
  Interventions: Drug: Selpercatinib
- 150 mg Ranitidine dosed with 160 mg Selpercatinib (Experimental): Participants received 150 mg ranitidine twice a day orally for 11 days (Study Days 8 to 18) with a single oral dose of 160 mg Selpercatinib (Study Day 12).
  Interventions: Drug: Selpercatinib; Drug: Ranitidine
- 40 mg Omeprazole dosed with 160 mg Selpercatinib (Experimental): Participants received 40 mg omeprazole once daily for 11 days (Study Days 19 to 29) with a single oral dose of 160 mg Selpercatinib (Study Day 23).
  Interventions: Drug: Selpercatinib; Drug: Omeprazole

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292
Drug: Ranitidine — Administered orally.
  Arms: 150 mg Ranitidine dosed with 160 mg Selpercatinib
Drug: Omeprazole — Administered orally.
  Arms: 40 mg Omeprazole dosed with 160 mg Selpercatinib

SUMMARY:
The main purpose of this study is to learn about how H2 antagonist (ranitidine) and proton pump inhibitor (PPI) (omeprazole) affect Selpercatinib in healthy participants. Information about safety and tolerability will be collected. The study will last up to about 9 weeks, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening
* Require treatment with inducers or inhibitors of cytochrome P450 (CYP) CYP3A within 14 days before the first dose of study drug through the end of Period 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a fixed sequence study where participants receive Selpercatinib in Period 1, Selpercatinib in combination with Ranitidine in Period 2, and Selpercatinib in combination with Omeprazole in Period 3.
Groups:
- 160 mg Selpercatinib: Participants received a single oral dose of 160 mg Selpercatinib (Study Day 1).
- 150 mg Ranitidine Dosed With 160 mg Selpercatinib: Participants received 150 mg ranitidine twice a day (BID) orally for 11 days (Study Days 8 to 18) with a single oral dose of 160 mg Selpercatinib (Study Day 12).
Period: Period 1 - Day 1 to Day 8
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Started | 20 | 0 | 0
Received at Least One Dose of Study Drug | 20 | 0 | 0
Completed | 20 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2 - Day 8 to Day 19
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Started | 0 (Participants were assigned to this arm only during Period 1.) | 20 | 0 (Participants were assigned to this arm only during Period 3.)
Completed | 0 | 17 | 0
Not Completed | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Period 3 - Day 19 to Day 29
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Started | 0 (Participants were assigned to this arm only during Period 1.) | 0 (Participants were assigned to this arm only during Period 2.) | 17
Completed | 0 | 0 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Study Participants: Participants received a single oral dose of 160 mg Selpercatinib (Study Day 1).
  Participants received 150 mg ranitidine twice a day orally for 11 days (Study Days 8 to 18) with a single oral dose of 160 mg Selpercatinib (Study Day 12).
  Participants received 40 mg omeprazole once daily for 11 days (Study Days 19 to 29) with a single oral dose of 160 mg Selpercatinib (Study Day 23).
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t of Selpercatinib. The analysis of variance (ANOVA) model was performed on the natural log (ln)-transformed PK parameters and included calculation of geometric least squares (LS) means and the difference between treatment geometric LS means, as well as their corresponding 90% confidence intervals (CIs). The ratios of geometric LS mean and 90% CI for the ratio of the PK parameter for each comparison was constructed using the exponentiation of the difference and the CIs from the ANOVA analyses.
Time Frame: PK: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 post Selpercatinib dose on Day 1 - Period 1, Day 12 - Period 2, and Day 23 - Period 3
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for AUC0-t.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter(h*ng/mL)
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 17 | 17
hour*nanograms per milliliter(h*ng/mL) | 21600 (31.4) | 19100 (31.9) | 21000 (27.4)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib vs 150 mg Ranitidine Dosed With 160 mg Selpercatinib; Fasted State; Test type: Superiority; ANOVA; Geometric Least Squares Mean (LSM) Ratio = 0.900, 90% CI 2-sided [0.797 to 1.02]
Statistical Analysis 2: Comparison: 160 mg Selpercatinib vs 40 mg Omeprazole Dosed With 160 mg Selpercatinib; Fed state; Test type: Superiority; ANOVA; Geometric LS Mean Ratio = 0.990, 90% CI 2-sided [0.876 to 1.12]

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib
Description: PK: AUC0-inf of Selpercatinib. The ANOVA model was performed on the natural log (ln)-transformed PK parameters and included calculation of geometric LS means and the difference between treatment geometric LS means, as well as their corresponding 90% CIs. The ratios of geometric LS mean and 90% CI for the ratio of the PK parameter for each comparison was constructed using the exponentiation of the difference and the CIs from the ANOVA analyses.
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for AUC0-inf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
h*ng/mL | 21800 (31.2) | 19900 (33.5) | 21100 (27.4)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib vs 150 mg Ranitidine Dosed With 160 mg Selpercatinib; Fasted state; Test type: Superiority; ANOVA; Geometric LS Mean Ratio = 0.932, 90% CI 2-sided [0.829 to 1.05]
Statistical Analysis 2: Comparison: 160 mg Selpercatinib vs 40 mg Omeprazole Dosed With 160 mg Selpercatinib; Fed State; Test type: Superiority; ANOVA; Geometric LS Mean Ratio = 1.00, 90% CI 2-sided [0.888 to 1.13]

3. Primary Outcome: PK: Percentage of Area Under the Plasma Concentration-Time Curve (AUC) That is Due to Extrapolation From Last Measurable Concentration to Infinity (%AUCextrap) of Selpercatinib
Description: PK: %AUCextrap of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for %AUCextrap.
Measure: Median (Full Range); unit: percentage of (%) of AUCextrap
Groups:
- 40 mg Omeprazole Dosed With 160mg Selpercatinib: Participants received 40 mg omeprazole once daily for 11 days (Study Days 19 to 29) with a single oral dose of 160 mg Selpercatinib (Study Day 23).
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
percentage of (%) of AUCextrap | 0.337 [0.136 to 3.00] | 0.818 [0.137 to 2.02] | 0.612 [0.103 to 1.59]

4. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib. The ANOVA model was performed on the natural log (ln)-transformed PK parameters and included calculation of geometric LS means and the difference between treatment geometric LS means, as well as their corresponding 90% CIs. The ratios of geometric LS mean and 90% CI for the ratio of the PK parameter for each comparison was constructed using the exponentiation of the difference and the CIs from the ANOVA analyses.
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
ng/mL | 1650 (58.4) | 1330 (67.8) | 1220 (63.4)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib vs 150 mg Ranitidine Dosed With 160 mg Selpercatinib; Fasted State; Test type: Superiority; ANOVA; Geometric LS Mean Ratio = 0.818, 90% CI 2-sided [0.680 to 0.985]
Statistical Analysis 2: Comparison: 160 mg Selpercatinib vs 40 mg Omeprazole Dosed With 160 mg Selpercatinib; Fed state; Test type: Superiority; ANOVA; Geometric LS Mean Ratio = 0.782, 90% CI 2-sided [0.645 to 0.949]

5. Primary Outcome: PK: Time of Maximum Observed Concentration (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for tmax.
Measure: Median (Full Range); unit: hour
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
hour | 2.00 [1.00 to 3.00] | 1.83 [1.00 to 24.00] | 3.00 [1.50 to 6.00]

6. Primary Outcome: PK: Apparent Volume of Distribution (Vz/F)
Description: PK: Vz/F of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
liter | 259 (44.2) | 331 (59.1) | 300 (48.6)

7. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Selpercatinib
Description: PK: CL/F of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 19 | 17
liter per hour (L/h) | 7.35 (31.2) | 8.03 (33.5) | 7.58 (27.4)

8. Primary Outcome: PK: Apparent Terminal Elimination Half-life (t½) of Selpercatinib
Description: PK: t½ of Selpercatinib
Time Frame: as for outcome 1
Population: All enrolled or randomized participants who received at least one dose of study drug with evaluable data for t½.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
Number analyzed (Participants) | 20 | 18 | 17
hour | 24.4 (35.4) | 29.3 (33.5) | 27.4 (30.1)

ADVERSE EVENTS:
Time Frame: Baseline through Day 37
Description: All enrolled or randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 160 mg Selpercatinib | 150 mg Ranitidine Dosed With 160 mg Selpercatinib | 40 mg Omeprazole Dosed With 160 mg Selpercatinib
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 5/20 | 11/20 | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 160 mg Selpercatinib (N=20) | 150 mg Ranitidine Dosed With 160 mg Selpercatinib (N=20) | 40 mg Omeprazole Dosed With 160 mg Selpercatinib (N=17)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/4 (0) | 1/4 (1) | 0/3 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/16 (1) | 0/16 (0) | 0/14 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT05338502/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT05338502/SAP_001.pdf